CLINICAL TRIAL: NCT03836547
Title: Feasibility of a Multi Component Intervention in Patients With Severe Dyspnea and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-001832
Record Dates: First submitted 2019-01-21; First posted 2019-02-11 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: COPD; Emphysema; Lung Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Lung Diseases

STUDY DESIGN:
Intervention Model Description: Patients with lung disease and a BMI of 35 or greater with significant shortness of breath will be randomized to a multicomponent intervention vs a wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent Intervention for weight loss (Experimental): 12-week intervention that consists of Weight Watcher on-line program, Garmin Fitness Tracker, blue-tooth scale, and telephonic health coaching.
  Interventions: Behavioral: Coaching and Weight Loss for patients with dyspnea
- Wait-list Control (Active Comparator): The participant will receive usual care for 12 weeks and then will compassionately be offered the active intervention.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Coaching and Weight Loss for patients with dyspnea — Patients with lung disease and a BMI of 35 or greater who suffer from shortness of breath will be invited to participate in a study involving a commercial weight loss application with health coaching. The patients will subscribe on their own to the weight loss application. The patients will be provided with a blue tooth scale so that they may weigh themselves weekly. A health coach will call them weekly for 8 weeks.
  Arms: Multicomponent Intervention for weight loss
Behavioral: Active Control — Participants will receive usual care for 12 weeks followed by the active intervention.
  Arms: Wait-list Control

SUMMARY:
Researchers are trying to test the effectiveness and feasibility of a multicomponent lifestyle intervention to support weight loss decreases dyspnea in obese people with chronic lung disease and clinically significant breathlessness.

DETAILED DESCRIPTION:
Patient will be randomized to a 12-week intervention that uses the Weight watchers lifestyle program online, a Garmin Fitness Tracker, blue tooth scale and receive health coaching vs a wait-list control group.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years.
* BMI >=35
* Dyspnea MRC class II or greater
* Diagnosis of lung disease
* Signed informed consent

Exclusion Criteria

* BMI <35
* Pregnancy
* Recent respiratory illness (within the last 6 weeks)
* Recent exacerbation of chronic lung disease (within the last 6 weeks)
* Already participating in a structured diet and/or exercise program
* Medical contraindication to weight loss (cancer)
* Medical contraindication to unsupervised exercise (unstable angina)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Breathlessness | baseline to 12 weeks
  Chronic Respiratory Questionnaire Dyspnea

SECONDARY OUTCOMES:
Lean Body Mass (lbs.)using InBody 770 Scale | baseline to 12 weeks
  InBody770 analyzer to define Lean Body Mass (total body weight minus weight of fat). This measure includes organs, skin, bones, water and muscle.
Skeletal Muscle Mass (lbs.) using InBody 770 Scale | baseline to 12 weeks
  InBody770 analyzer to define skeletal muscle mass (total weight of muscle)
Percent Body Fat using InBody 770 Scale | baseline to 12 weeks
  InBody770 analyzer to define percent body fat
Weight using InBody 770 Scale | baseline to 12 weeks
  InBody770 analyzer to define weight
Body Mass Index using InBody 770 Scale | baseline to 12 weeks
  InBody770 analyzer to define Body Mass Index (BMI) is weight in kilograms divided by height in meters squared. A BMI of 25 or below is considered healthy.
Mindful Eating | baseline to 12 weeks
  Mindful Eating Questionnaire- 28 item instrument with a score range of 1-4. Higher scores are associated with lower body mass indexes.
Daily Steps | baseline to 12 weeks
  Number of steps participant takes in a day recorded by Actigraph Activity tracker.
Daily Sedentary Time | baseline to 12 weeks
  Actigraph Activity Tracker to determine the amount of time (minutes) spend sedentary status
Daily Physical Activity | baseline to 12 weeks
  Actigraph Activity Tracker to define the amount of time spent in mild to moderate and vigorous physical activity define by METs
Exercise Capacity | baseline to 12 weeks
  Six-Minute Walking Test
Sleep Time Measures | baseline to 12 weeks
  Actigraph to measure total sleep time
Sleep Efficiency | baseline to 12 weeks
  Time sleeping/ Time reclined
Disease specific quality of life | baseline to 12 weeks
  Chronic Respiratory Questionnaire measures Fatigue , Emotions and Mastery and is a 20 item questionnaire with a range of 1-7. A higher score is best.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials